CLINICAL TRIAL: NCT06111235
Title: A Phase 3, Randomized Study of Adjuvant Cretostimogene Grenadenorepvec Versus Observation for the Treatment of Intermediate Risk Non-Muscle Invasive Bladder Cancer (IR-NMIBC) Following Transurethral Resection of Bladder Tumor (TURBT)
Brief Title: A Study of Adjuvant Cretostimogene Grenadenorepvec for Treatment of Intermediate Risk NMIBC Following TURBT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIVOT-006
Record Dates: First submitted 2023-10-25; First posted 2023-11-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non Muscle Invasive Bladder Cancer; Urologic Cancer; Bladder Cancer; Urothelial Carcinoma
Keywords: Urology; Bladder Cancer; Non Muscle Invasive Bladder Cancer; Intermediate Risk Non Muscle Invasive Bladder Cancer; Cretostimogene Grenadenorepvec
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urologic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — dodecyl maltoside

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, open-label, randomized trial designed to evaluate the RFS of TURBT followed by adjuvant cretostimogene versus TURBT alone for the treatment of participants with IR-NMIBC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cretostimogene after TURBT (Experimental): Following screening confirmation of IR-NMIBC and complete resection of the tumor, participants will be treated with adjuvant cretostimogene.
  Interventions: Drug: Cretostimogene Grenadenorepvec; Other: n-dodecyl-B-D-maltoside
- Observation after TURBT (No Intervention): Following screening confirmation of IR-NMIBC and complete resection of tumor, participants will enter surveillance.
  Participants who recur with IR-NMIBC after TURBT and surveillance will be offered treatment with cretostimogene as per the treatment schedule in Arm A. This arm will be called the Extension Arm.

INTERVENTIONS:
Drug: Cretostimogene Grenadenorepvec — Engineered Oncolytic Adenovirus
  Other Names: CG0070
  Arms: Cretostimogene after TURBT
Other: n-dodecyl-B-D-maltoside — Transduction-enhancing agent
  Other Names: DDM
  Arms: Cretostimogene after TURBT

SUMMARY:
This is a Phase 3, open-label, randomized trial designed to evaluate the RFS of TURBT followed by cretostimogene grenadenorepvec versus TURBT followed by surveillance for the treatment of participants with IR-NMIBC.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to cretostimogene grenadenorepvec after TURBT (Arm A) vs surveillance after TURBT (Arm B).

Participants in Arm A will receive an induction course and then quarterly maintenance courses of cretostimogene through Month 13, if there is no disease recurrence.

Disease status will be assessed using urine cytology, cystoscopy, and directed TURBT/biopsy (if indicated) every 3 months for the first 2 years after randomization and then every 6 months for an additional year or until disease recurrence. CT Urogram/MRU every 12 months.

Participants in Arm B who recur with IR-NMIBC after TURBT and surveillance will be offered treatment with cretostimogene as per the treatment schedule in Arm A.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed IR-NMIBC, per American Urologic Association/Society of Urologic Oncology/National Comprehensive Cancer Network guidelines, within 90 days of participant randomization:

  1. Recurrent LG Ta within 12 months of prior LG or HG (HG Ta ≤ 3 cm) tumor
  2. Solitary LG Ta >3 cm tumor
  3. Multifocal LG Ta tumors
  4. Primary and solitary HG Ta ≤3 cm tumor
  5. LG T1 tumor
* All visible disease removed by TURBT within 90 days of study randomization
* Acceptable baseline organ function

Exclusion Criteria:

* High-risk NMIBC (e.g., HG T1, Recurrent or multifocal HG Ta>3cm tumor(s), CIS)
* Low-Risk NMIBC (e.g., solitary LG Ta ≤3 cm tumor)
* Disease in the prostatic urethra at any time or in the upper genitourinary tract within 24 months of randomization
* Muscle-invasive bladder cancer, locally advanced or metastatic bladder cancer
* Prior treatment with any human adenovirus serotype 5 based therapy (e.g., Adstiladrin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) | 29 months
  Recurrence free survival (RFS) of cretostimogene after TURBT versus surveillance after TURBT

SECONDARY OUTCOMES:
Recurrence Free Survival (RFS) at 6 months, 12 months and 24 months | 27 months (RFS at 6 months), 33 months (RFS at 12 months) and 45 months (RFS at 24 months)
  Recurrence free survival (RFS) of cretostimogene after TURBT versus surveillance after TURBT at 12 months and 24 months
Incidence of Adverse Events | 34 months
  Safety of cretostimogene following TURBT

CONTACTS AND LOCATIONS:
Overall Officials: Max Kates, MD, Principal Investigator — Johns Hopkins University
Locations (95):
- United States (90):
  - Urology Centers of Alabama PC, Homewood, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Institute of Urology PLLC, Tucson, Arizona
  - Arkansas Urology PA, Little Rock, Arkansas
  - Michael G. Oefelein MD Clinical Trials, Bakersfield, California
  - USC/Keck Department of Urology, Los Angeles, California
  - Tower Urology, Los Angeles, California
  - Sun Kim Urology, Orange, California
  - University of California Irvine Medical Center (UCIMC), Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Stanford University School of Medicine, Stanford, California
  - Colorado Clinical Research, Aurora, Colorado
  - Urology Associates, PC, Lone Tree, Colorado
  - Hartford HealthCare Medical Group, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advanced Urology Institute, Daytona Beach, Florida
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Lakeland Regional Health, Lakeland, Florida
  - Advanced Urology Institute, LLC, Largo, Florida
  - University of Miami, Miami, Florida
  - Emory Winship Cancer Center, Atlanta, Georgia
  - Velocity Clinical Research- Savanah Urological Associates, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - UroPartners LLC, Glenview, Illinois
  - Duly Health and Care, Lisle, Illinois
  - Urology of Indiana, LLC, Carmel, Indiana
  - Urology of Indiana, Greenwood, Indiana
  - Urology Center of Iowa Research, West Des Moines, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Wichita Urology Group, Wichita, Kansas
  - First Urology, PSC, Louisville, Kentucky
  - Southern Urology, Lafayette, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Associates, LLC, Baltimore, Maryland
  - Johns Hopkins Hospital Green Spring Station, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cancer Center at Beth Israel Deaconess Medical Center - Research, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Urology, Roseville, Michigan
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Urology Group, Southaven, Mississippi
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Urology Nevada, Reno, Nevada
  - Garden State Urology, LLC- Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey - Cancer Center, New Brunswick, New Jersey
  - Integrated Medical Professionals PLLC, New York, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Cancer Center, Durham, North Carolina
  - Urology Group, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Oregon Urology Insititute, Springfield, Oregon
  - Midlantic Urology, Bala-Cynwyd, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Lowcountry Urology Clinics, North Charleston, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Urology Associates, P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Amarillo Urology Research, LLC, Amarillo, Texas
  - Urology Associates of North Texas, Arlington, Texas
  - Urology Austin, PLLC, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio PA, San Antonio, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah- Huntsman Cancer Institute, Salt Lake City, Utah
  - Urology of Virginia (UVA) - Virginia Beach (Devine-Tidewater Urology), Virginia Beach, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Spokane Urology- Southside, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - University of Wisconsin Medical Foundation, Madison, Wisconsin
- Canada (5):
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Nova Scotia Health Centre of Applied Urology Research, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - University Health Network (UHN) - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Center - Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang SS, Boorjian SA, Chou R, Clark PE, Daneshmand S, Konety BR, Pruthi R, Quale DZ, Ritch CR, Seigne JD, Skinner EC, Smith ND, McKiernan JM. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline. J Urol. 2016 Oct;196(4):1021-9. doi: 10.1016/j.juro.2016.06.049. Epub 2016 Jun 16. PMID 27317986
- See also: NCCN Guidelines Bladder Cancer 3.2023 — https://www.nccn.org/guidelines/recently-published-guidelines